CLINICAL TRIAL: NCT02642302
Title: Can The Rest Interval Time Provide Superior Gains on VO2max, Aerobic and Anaerobic Performance Obtained With High Intensity Interval Training (HIIT)? a Randomized Controlled Study
Brief Title: Rest Time on Gain Aerobic and Anaerobic Performance
Acronym: Performance
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidade Federal do Rio de Janeiro (Other)
Responsible Party: Principal Investigator, Alberto Souza de Sá Filho, Doctorade in Mental Health, Universidade Federal do Rio de Janeiro
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: UNIVERSO-02
Record Dates: First submitted 2015-12-05; First posted 2015-12-30 (Estimated); Last update posted 2015-12-30 (Estimated); Status verified 2015-12

CONDITIONS: Healthy
Keywords: VO2Max; Aerobic Exercise; Physical Conditioning
MeSH Terms: conditions — Motor Activity | interventions — RE1-silencing transcription factor; High-Intensity Interval Training

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- HIIT With 60 sec Rest (Experimental): The experimental (1) group will be submitted at Six reps of 30 seconds of high intensity interval training (all out) with 60 seconds of interval rest for a total of 30 sessions of training. Dependents variables such as VO2Max and performance parameters are estimated before and after training sessions
  Interventions: Behavioral: HIIT With120 sec Rest
- HIIT With 120 sec Rest (Experimental): The experimental (2) group will be submitted at Six reps of 30 seconds of high intensity interval training (all out) with 120 seconds of interval rest for a total of 30 sessions of training. Dependents variables such as VO2Max and performance parameters are estimated before and after training sessions
  Interventions: Behavioral: HIIT With 60 sec Rest
- Control (Active Comparator): Continuous exercise at 50-55% of VO2max with similar total work
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: HIIT With 60 sec Rest — 30 sessions of High intensity interval training (all out) with 30 seconds of stimulous with 60 seconds rest on VO2Max and aerobic/ anaerobic performance
  Other Names: High intensity interval training with 60 seconds rest; HIIT
  Arms: HIIT With 120 sec Rest
Behavioral: HIIT With120 sec Rest — 30 sessions of High intensity interval training (all out) with 30 seconds of stimulous with 120 seconds rest on VO2Max and aerobic/ anaerobic performance
  Other Names: High intensity interval training with 120 seconds rest
  Arms: HIIT With 60 sec Rest
Behavioral: Control — Continuous exercise at 50-55% VO2Max with similar total work of interval training
  Other Names: Control Continuous Exercise
  Arms: Control

SUMMARY:
Based on studies of high intensity interval training (HIIT) in the literature, higher gains in VO2max and performance are obtained in short periods of training time. However, different designs training configurations, for example, changing the time interval, could influence such gains on VO2max and aerobic performance. The aim of the study was to observe the possible influences of diferetes types of rest intervals in high intensity interval exercise protocol on VO2max, and the aerobic and anaerobic performances in 12 weeks of training.

DETAILED DESCRIPTION:
12-week experiment will be conducted, with a total of 30 high intensity interval training (HIIT) sessions in cycle ergometer. Both the first and the last week will serve to stabilize the basic values and also repeated after training. So, every other day will be held: 1) risk stratification for coronary artery disease, anthropometric measurements, cardiopulmonary test maximum effort; 2) stabilization of cardiopulmonary test values, determining the aerobic dependent variables: VO2max, peak power - PP, occurrence of power VO2max - PVO2Máx, maximum heart rate - HRMax, as well as familiarization with the HIIT protocol; 3) anaerobic performance test of 30 seconds determining the anaerobic dependent variables: peak lactate - LA, anaerobic power peak - PP, average power - PM. After the dependent variables have established, the subjects will be randomly distributed among three groups: two experimental and one control, and subjected to 30 sessions of HIIT (all out)with 30 seconds of stimulation in cycle ergometer, differentiated only by the recovery time (60 seconds and 120 seconds). The control group had only one continuous aerobic exercise (50-55% VO2max) with an average time similar to other training.

ELIGIBILITY:
Inclusion Criteria:

* practitioners of aerobic activities for 6 mounths
* negative prognosis for cardiovascular or metabolic disease

Exclusion Criteria:

* muscle injuries
* use ergogenic resources
* cardiovascular disease
* other limitations

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2015-12; Primary Completion 2016-02 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
Oxygen Intake (VO2Max) Against of Differents Rest Time of High Intensity Interval Training | Change From Baseline VO2Max after 12 Weeks of High Intensity Interval Training

SECONDARY OUTCOMES:
Aerobic and Anaerobic Power Peak Performance Against of Differents Rest Time of High Intensity | Change From Baseline in Aerobic and Anaerobic Performance after 12 Weeks of High Intensity Interval Training
Lactate Concentration | Change From Baseline in Lactate Concentration after 12 Weeks of High Intensity Interval Training

CONTACTS AND LOCATIONS:
Overall Officials: Sérgio Machado, PhD, Study Director — Salgado de Oliveira University